CLINICAL TRIAL: NCT02965729
Title: Our Lifestyles, Our Lives: Obesity Treatment and Physical Activity Promotion for Underserved Children and Adolescents
Brief Title: Our Lifestyles Our Lives
Acronym: OLOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Our Lady of the Lake Hospital (Other); American Council on Exercise (Other)
Responsible Party: Principal Investigator, Amanda Staiano, Assistant Professor - Research, Pennington Biomedical Research Center
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 2014-012
Record Dates: First submitted 2016-11-14; First posted 2016-11-17 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Pediatric Obesity; Weight Loss
Keywords: behavior goals; self-monitoring; pedometer; physical activity
MeSH Terms: conditions — Pediatric Obesity; Weight Loss; Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Pedometer (Active Comparator): Participants only participated in the family-based weight management intervention. Participants were not given a pedometer or step goals.
  Interventions: Behavioral: Family-based weight management
- Pedometer Only (Active Comparator): In addition to participating in the family-based weight management intervention, participants were given a pedometer and instructions at session 1. Participants were asked to wear the pedometer every day for the entirety of the program and return at session 10. No step goals were provided.
  Interventions: Behavioral: Family-based weight management; Behavioral: Pedometer
- Pedometer Plus Step Goals (Active Comparator): In addition to participating in the family-based weight management intervention, participants were given a pedometer and instructions at session 1. Participants were asked to wear the pedometer every day for the entirety of the program and return at session 10. Participants were given individualized step goals to increase their activity by 500 steps each week (above baseline calculated as average daily steps/day during week 1).
  Interventions: Behavioral: Family-based weight management; Behavioral: Pedometer; Behavioral: Individualized step goals

INTERVENTIONS:
Behavioral: Family-based weight management — The "Our Lifestyles, Our Lives" family-based weight management intervention consisted of 10 weekly 90-minute group sessions focused on physical activity, nutrition, and behavioral modification. Parents and siblings were encouraged to join the participant in these sessions. Sessions were interactive and included cooking demonstrations, light to moderate intensity physical activity that engaged all family members, and behavioral counseling sessions in both mixed (parent and child) and parent-only format.
Behavioral: Pedometer — In addition to participating in the family-based weight management intervention, participants were given a pedometer (Omron HJ-324U, Omron Healthcare, Lake Forest, IL) and instructions at session 1. Participants were asked to wear the pedometer every day for the entirety of the program and return at session 10.
  Other Names: Activity monitor
  Arms: Pedometer Only; Pedometer Plus Step Goals
Behavioral: Individualized step goals — In addition to participating in the family-based weight management intervention, participants were given a step goal to increase their activity by 500 steps each week (above baseline calculated as average daily steps/day during week 1).
  Arms: Pedometer Plus Step Goals

SUMMARY:
The purpose of the study was to examine the influence of step goals with pedometers to improve children's weight loss, physical activity, and psychosocial health during behavioral treatment. Children with overweight or obesity were assigned to receive the behavioral treatment alone, plus pedometers, or plus pedometers with step goals.

DETAILED DESCRIPTION:
A total of 105 overweight and obese children ages 8 to 17 years participated in a 10-week family-based weight management intervention focusing on physical activity, nutrition, and behavioral modification. A quasi-experimental design was used to group cohorts into three conditions: two cohorts had no pedometer (n=24); two cohorts had pedometer only (n=25); and four cohorts had pedometer with step goals (i.e. 500 steps/day weekly increase above baseline; n=56). Height and weight were measured at baseline and week 10 and used to calculate body mass index (BMI). Analysis of covariance was performed to examine difference by condition for change in weight, BMI, and BMI z-score, controlling for age and baseline value. Differences in steps/day and psychosocial health were compared between the two pedometer conditions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8-17 years old
* BMI ≥ 95th percentile or have a BMI ≥ 85th percentile with comorbidities (e.g. hypertension, heart disease, type 2 diabetes, insulin resistance, sleep apnea, orthopedic problems, or fatty liver disease)

Exclusion Criteria:

* None.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Staiano, PhD, Principal Investigator — Pennington Biomedical Research Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Staiano AE, Beyl RA, Hsia DS, Jarrell AR, Katzmarzyk PT, Mantzor S, Newton RL Jr, Tyson P. Step Tracking with Goals Increases Children's Weight Loss in Behavioral Intervention. Child Obes. 2017 Aug;13(4):283-290. doi: 10.1089/chi.2017.0047. Epub 2017 Apr 25. PMID 28440662

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Pedometer | Pedometer Only | Pedometer Plus Step Goals
Started | 24 | 25 | 56
Completed | 17 | 22 | 45
Not Completed | 7 | 3 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Pedometer | Pedometer Only | Pedometer Plus Step Goals | Total
Number analyzed (Participants) | 24 | 25 | 56 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 25 | 56 | 105
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (2.5) | 11.7 (2.1) | 13.1 (2.6) | 12.4 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 39 | 73
  Male | 6 | 9 | 17 | 32
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 56 | 105

OUTCOME MEASURES:

1. Primary Outcome: BMI Z-score Change
Description: Height was measured at sessions 1 and 10 using a stadiometer. Weight was measured at each session using a calibrated scale. BMI z-score was calculated from the Centers for Disease Control and Prevention macro program based on the sex, height, and age of the child. Change was calculated as difference between baseline and end of 10-week study.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | No Pedometer | Pedometer Only | Pedometer Plus Step Goals
Number analyzed (Participants) | 17 | 22 | 45
z score | 0.01 (0.04) | -0.03 (0.04) | -0.03 (0.05)

2. Secondary Outcome: BMI Change
Description: BMI was calculated as weight in kg divided by height in meters squared. Change was calculated as difference between baseline and end of 10-week study.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | No Pedometer | Pedometer Only | Pedometer Plus Step Goals
Number analyzed (Participants) | 17 | 22 | 45
kg/m2 | 0.43 (0.82) | -0.24 (0.78) | -0.37 (0.92)

3. Secondary Outcome: Body Weight Change
Description: Weight was measured using a calibrated scale. Change was calculated as difference between baseline and end of 10-week study.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | No Pedometer | Pedometer Only | Pedometer Plus Step Goals
Number analyzed (Participants) | 17 | 22 | 45
kg | 1.12 (1.9) | 0.23 (1.87) | -0.49 (2.06)

4. Secondary Outcome: Quality of Life Kidscreen-10 Index Change
Description: Health-related quality of life was measured using the Kidscreen-10 Index. Change was calculated as difference between baseline and end of 10-week study. the scale ranged from 0 to 15, with higher values indicating a better outcome.
Time Frame: 10 weeks
Population: Data were not collected for the ''No Pedometer'' cohorts.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Pedometer | Pedometer Only | Pedometer Plus Step Goals
Number analyzed (Participants) | 0 | 20 | 39
units on a scale |  | 2.2 (4.5) | 0.9 (5.3)

5. Secondary Outcome: Physical Activity Enjoyment Change
Description: Physical activity enjoyment was measured using the Physical Activity Enjoyment Scale (PACES). Change was calculated as difference between baseline and end of 10-week study. The scale ranged from 0 to 32, with higher values indicating a better outcome.
Time Frame: 10 weeks
Population: Data were not collected for the ''No Pedometer'' cohorts.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Pedometer | Pedometer Only | Pedometer Plus Step Goals
Number analyzed (Participants) | 0 | 20 | 39
units on a scale |  | 0.02 (8.25) | 2.66 (10.9)

6. Secondary Outcome: Subjective Health Change
Description: Subjective health was measured using a 1-item Likert scale ("In general, how would you say your health is?"). Change was calculated as difference between baseline and end of 10-week study. The scale ranged from 0 to 4, with higher values indicating a better outcome.
Time Frame: 10 weeks
Population: Data were not collected for the ''No Pedometer'' cohorts.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Pedometer | Pedometer Only | Pedometer Plus Step Goals
Number analyzed (Participants) | 0 | 20 | 39
units on a scale |  | 0.55 (1.34) | 0.66 (1.00)

7. Secondary Outcome: Physical Activity Change
Description: Physical activity was measured in the pedometer only and pedometer plus goals groups using an Omron pedometer (Omron HJ-324U, Omron Healthcare, Lake Forest, IL). Change was calculated as difference between baseline and end of 10-week study.
Time Frame: 10 weeks
Population: Pedometers were not worn in the "No Pedometer" cohorts and so data were not collected.
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | No Pedometer | Pedometer Only | Pedometer Plus Step Goals
Number analyzed (Participants) | 0 | 22 | 45
steps |  | -162 (620) | 1185 (425)

ADVERSE EVENTS:
Arm/Group | No Pedometer | Pedometer Only | Pedometer Plus Step Goals
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 0/56
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes